CLINICAL TRIAL: NCT00762073
Title: Oral Viscous Budesonide Suspension (MB-7) in Subjects With Eosinophilic Esophagitis: A Randomized, Placebo-Controlled, Dose-Ranging Study in Children and Adolescents
Brief Title: Dose-Ranging Study of Oral Viscous Budesonide in Pediatrics With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPI-101-01
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): Low Dose Group
  Interventions: Drug: budesonide
- 3 (Experimental): Medium Dose Group
  Interventions: Drug: budesonide
- 4 (Experimental): High Dose Group
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — oral suspension
  Arms: 2; 3; 4
Drug: placebo — oral suspension matching budesonide
  Arms: 1

SUMMARY:
This is a randomized, placebo-controlled, parallel-arm, dose-ranging study in subjects with eosinophilic esophagitis, 2-18 years of age. Eligible subjects will be randomized into one of four treatment groups. The Treatment Period will be 12 weeks during which subjects will visit the clinic at study weeks 0 (Baseline Visit), 2, 4, 8 and 12 (Final Treatment Evaluation) for clinical symptom assessment and safety evaluation (including adverse events and vital signs). All study treatments (active drug and placebo) will be administered orally twice daily during the Treatment Period, once in the morning after breakfast and once in the evening at bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 2-18 years, inclusive
* History of clinical symptoms of esophageal dysfunction intermittently or continuously
* Histologic evidence of EoE with a peak eosinophil count of greater than or equal to 20 eosinophils per HPF, from two or more levels of the esophagus, within six weeks prior to the Baseline Visit
* At the Baseline Visit, subjects must have symptoms with a total EoE Clinical Symptom Score of greater than or equal to 3
* Willingness and ability to continue the dietary therapy, environmental therapy, and/or medical regimens (including gastric acid suppression, if any) in effect at the Screening Visit
* Females of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin) prior to randomization into the study and sexually active subjects must agree to continue acceptable birth control measures throughout the duration of the study
* Written informed consent (parent or legal guardian) and, as appropriate, subject assent

Exclusion Criteria:

* Current use of immunomodulatory therapy (or anticipated use within 12 weeks following the Baseline Visit)
* Diagnosis of inflammatory bowel disease
* Chronic viral infection or immunodeficiency condition (current)
* Use of swallowed topical corticosteroids for EoE in the 1 month prior to the biopsy required for entrance to this study or at any time between the biopsy and the Baseline Visit
* Use of systemic (oral or parenteral) corticosteroid within 1 month prior to the biopsy required for entrance to this study or at any time between the biopsy and the Baseline Visit
* Morning plasma cortisol level below the lower limit of normal (per Central Laboratory reference range) at the Screening Visit
* Upper gastrointestinal bleeding within 1 month prior to the Screening Visit or between the Screening Visit and Baseline Visit
* Current use of anticoagulants
* Current disease of the gastrointestinal tract aside from the current EoE diagnosis
* Evidence of concurrent eosinophilic gastritis, enteritis, colitis, or proctitis
* Evidence of active infection with Helicobacter pylori
* Evidence of unstable asthma or changes in asthma or allergic rhinitis therapy within 1 month prior to the biopsy required for entrance to this study
* Any female who is pregnant, who is planning to become pregnant, or who is breast-feeding
* Current evidence or history of hypersensitivity or idiosyncratic reaction to budesonide or any other ingredients of the study medication
* Current evidence of oropharyngeal or esophageal candidiasis
* Receipt of an investigational drug within 30 days prior to the biopsy required for entrance to this study
* Any condition or abnormality that, in the opinion of the Principal Investigator, would compromise the safety of the subject or successful conduct of the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2009-01-08 (Actual); Primary Completion 2010-04-02 (Actual); Study Completion 2010-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- United States (20):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - The Children's Hospital, Aurora, Colorado
  - Emory University-Emory Children's Center, Atlanta, Georgia
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Center for Children's Digestive Health, Park Ridge, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - The Center for Human Nutrition, Omaha, Nebraska
  - Pediatric Gastroenterology and Nutrition Associates, Las Vegas, Nevada
  - South Jersey Pediatric Gastroenterology, Mays Landing, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Center for Digestive Health, Greenville, South Carolina
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Medical College of Virginia, Richmond, Virginia
  - Carilion Pediatric Gastroenterology, Roanoke, Virginia

REFERENCES:
- [Derived] Gupta SK, Hill M, Vitanza JM, Farber RH, Desai NK, Williams J, Song IH. Pharmacokinetics of Budesonide Oral Suspension in Children and Adolescents With Eosinophilic Esophagitis. J Pediatr Gastroenterol Nutr. 2022 Aug 1;75(2):186-191. doi: 10.1097/MPG.0000000000003482. Epub 2022 Jun 6. PMID 35666852
- [Derived] Gupta SK, Vitanza JM, Collins MH. Efficacy and safety of oral budesonide suspension in pediatric patients with eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2015 Jan;13(1):66-76.e3. doi: 10.1016/j.cgh.2014.05.021. Epub 2014 Jun 4. PMID 24907502

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo twice daily at bedtime (hs) and after breakfast (qAM, pc) for 12 weeks with a 3 week taper period.
- Low Dose: Participants received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc) for 12 weeks, with a total daily dose of 0.35 mg (2 to 9 years) or 0.50 mg (10 to 18 years), followed by a 3 week taper period.
- Medium Dose: Participants received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc) for 12 weeks, with a total daily dose of 1.4 mg (2 to 9 years) or 2.0 mg (10 to 18 years), followed by a 3 week taper period.
- High Dose: Participants received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and after breakfast (qAM, pc) for 12 weeks, with a total daily dose of 2.8 mg (2 to 9 years) or 4.0 mg (10 to 18 years), followed by a 3 week taper period.
Period: Overall Study
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Started | 21 | 21 | 20 | 20
Completed | 17 | 17 | 18 (One participant was enrolled and randomized then withdrew consent and did not receive study drug.) | 17
Not Completed | 4 | 4 | 2 | 3
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Significant Subject Noncompliance | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1
Not completed — Not on treatment for >/= 77 days | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set, defined as all randomized participants who received at least one dose of double-blind study drug. Treatment group assignment was the treatment actually received. One participant in the medium dose group was enrolled and randomized then withdrew consent and did not receive study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose | Total
Number analyzed (Participants) | 21 | 21 | 19 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (4.36) | 9.0 (5.88) | 10.2 (4.89) | 8.1 (4.58) | 9.1 (4.93)
Age, Customized [Count of Participants; unit: Participants]
  2 to 9 years | 12 | 12 | 10 | 12 | 46
  10 to 18 years | 9 | 9 | 9 | 8 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 4 | 15
  Male | 16 | 17 | 17 | 16 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Responded to Therapy
Description: Response was defined as a ≥50% reduction from baseline in the eosinophilic esophagitis (EoE) clinical symptom score (CSS) and a reduction in peak eosinophil count to ≤6/high power field (light microscopy) from esophageal biopsies collected at the final evaluation. The EoE CSS, scored from 0 to 18 by a doctor, assessed 6 categories: 1) heartburn, 2) abdominal pain, 3) nocturnal awakening with symptoms, 4) nausea, regurgitation, or vomiting, 5) anorexia or early satiety, and 6) dysphagia, odynophagia, or food impaction (a severe symptom). Each domain was scored as follows, based on symptoms in the 2 weeks prior to the assessment: 0 = No symptoms and no coping behaviors required; 1 = Mild: Symptoms limited to 1-3 days or no symptoms because coping behaviors were required to avoid symptoms; 2 = Moderate: Symptoms on >3 days, with or without minor coping behaviors; 3 = Severe: Symptoms interfered with activities of daily living or symptoms persisted and required major coping behaviors.
Time Frame: 12 weeks after the start of treatment
Population: The Full Analysis Set (FAS), defined as participants who received at least one dose of study drug and had evaluable post-baseline esophageal biopsy and clinical symptom data.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo twice daily at bedtime (hs) and after breakfast (qAM, pc) for 12 weeks, followed by a 3 week taper period.
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percentage of participants | 5.6 | 11.8 | 52.6 | 47.1
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.5282, Regression, Logistic — p-values comparing each active treatment group to placebo were determined by a logistic regression analysis with treatment (all four groups) and age as main effects; Odds Ratio (OR) = 2.239
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.0092, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 18.860
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.0174, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 15.009

2. Secondary Outcome: Percent of Participants With Histologic Response
Description: Histologic response was defined as a maximum peak eosinophil count at the final treatment evaluation of ≤6 eosinophils/high power field (light microscopy). The maximum peak was identified by examining the peak eosinophil counts obtained from the proximal, mid, and distal esophageal biopsies and selecting the maximum value.
Time Frame: 12 weeks after the start of treatment
Population: The FAS, defined as participants who received at least one dose of study drug and had evaluable post-baseline esophageal biopsy and clinical symptom data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percentage of participants | 5.6 | 23.5 | 52.6 | 94.1
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.1786, Regression, Logistic — p-values were determined by a logistic regression analysis with treatment (all four groups) and age group as main effects
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.0090, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percent of Participants With Histologic Remission
Description: Histologic remission was defined as a maximum peak eosinophil count at the final treatment evaluation of ≤1 eosinophils/high power field (light microscopy). The maximum peak was identified by examining the peak eosinophil counts obtained from the proximal, mid, and distal esophageal biopsies and selecting the maximum value.
Time Frame: 12 weeks after the start of treatment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percentage of participants | 0.0 | 11.8 | 42.1 | 76.5
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.4959, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.0040, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in Peak Eosinophil Count
Description: The maximum peak number of eosinophils at baseline and at the final treatment evaluation was identified by examining the peak eosinophil counts obtained from the proximal, mid, and distal esophageal biopsies and selecting the maximum value. A negative change from baseline indicates that eosinophil count has decreased.
Time Frame: Baseline, 12 weeks after the start of treatment
Population: The FAS, defined as all participants who received at least one dose of study drug and had evaluable post-baseline esophageal biopsy and clinical symptom data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percent change | 7.93 (84.162) | -52.62 (51.22) | -44.02 (89.106) | -94.75 (19.615)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0108, ANCOVA — p-values comparing percent change from baseline for each active treatment group to placebo were determined by an ANCOVA model with treatment and age strata as main effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.0208, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Endoscopy Score
Description: Esophageal endoscopy was used to assess the level of inflammation and eosinophilia. Four categories of endoscopic findings were evaluated and scored for this study: (1) pallor and diminished vascular markings; (2) furrowing with thickened mucosa; (3) presence of white mucosal plaques; and (4) concentric rings or strictures. For each category, 0 points were allocated if no esophageal sites were involved, 1 point if 1 or 2 esophageal sites were involved, and 2 points for pan-esophageal involvement (see Aceves et al., 2007). The maximum possible endoscopy score was 8 points. A negative change from baseline indicates that esophageal inflammation decreased.
Time Frame: Baseline, 12 weeks after the start of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
scores on a scale | -0.6 (2.28) | -0.9 (1.90) | -1.3 (2.23) | -2.2 (1.81)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.1095, ANCOVA — p-values comparing each active treatment group to placebo were determined by an ANCOVA model with treatment and age strata as main effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.0264, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percent of Participants With Clinical Response
Description: Response was defined as a ≥50% reduction from baseline in the eosinophilic esophagitis (EoE) clinical symptom score (CSS). The EoE CSS, scored from 0 to 18 by a doctor, assessed 6 categories: 1) heartburn, 2) abdominal pain, 3) nocturnal awakening with symptoms, 4) nausea, regurgitation, or vomiting, 5) anorexia or early satiety, and 6) dysphagia, odynophagia, or food impaction (a severe symptom). Each domain was scored as follows, based on symptoms in the 2 weeks prior to the assessment: 0 = No symptoms and no coping behaviors required; 1 = Mild: Symptoms limited to 1-3 days or no symptoms because coping behaviors were required to avoid symptoms; 2 = Moderate: Symptoms on >3 days, with or without minor coping behaviors; 3 = Severe: Symptoms interfered with activities of daily living or symptoms persisted and required major coping behaviors.
Time Frame: 12 weeks after the start of treatment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percentage of participants | 77.8 | 64.7 | 78.9 | 52.9
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.3769, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.9363, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.1235, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percent of Participants With Clinical Remission
Description: Clinical remission was defined as an eosinophilic esophagitis (EoE) clinical symptom score (CSS) of zero. EoE CSS, scored from 0 to 18 by a doctor, assessed 6 categories: 1) heartburn, 2) abdominal pain, 3) nocturnal awakening with symptoms, 4) nausea, regurgitation, or vomiting, 5) anorexia or early satiety, and 6) dysphagia, odynophagia, or food impaction (a severe symptom). Each domain was scored as follows, based on symptoms in the 2 weeks prior to the assessment: 0 = No symptoms and no coping behaviors required; 1 = Mild: Symptoms limited to 1-3 days or no symptoms because coping behaviors were required to avoid symptoms; 2 = Moderate: Symptoms on >3 days, with or without minor coping behaviors; 3 = Severe: Symptoms interfered with activities of daily living or symptoms persisted and required major coping behaviors.
Time Frame: 12 weeks after the start of treatment
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percentage of participants | 33.3 | 17.6 | 31.6 | 17.6
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.3444, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.9258, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.3215, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percent Change From Baseline in Eosinophilic Esophagitis (EoE) Clinical Symptom Score (CSS)
Description: The EoE CSS, scored from 0 to 18 by a doctor, assessed 6 categories: 1) heartburn, 2) abdominal pain, 3) nocturnal awakening with symptoms, 4) nausea, regurgitation, or vomiting, 5) anorexia or early satiety, and 6) dysphagia, odynophagia, or food impaction (a severe symptom). Each domain was scored as follows, based on symptoms in the 2 weeks prior to the assessment: 0 = No symptoms and no coping behaviors required; 1= Mild: Symptoms limited to 1-3 days or no symptoms because coping behaviors were required to avoid symptoms; 2= Moderate: Symptoms on >3 days, with or without minor coping behaviors; 3= Severe: Symptoms interfered with activities of daily living or symptoms persisted and required major coping behaviors. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, 12 weeks after the start of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 17
percent change | -64.46 (45.759) | -60.83 (30.347) | -65.89 (32.382) | -47.21 (40.790)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.6729, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.8894, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.1532, ANCOVA — [p-value comment as in outcome 4, analysis 1]

9. Secondary Outcome: Change From Baseline in Physician's Global Assessment Score of Disease Severity
Description: Physician investigators were asked to complete a visual analog scale (VAS) to provide a global assessment of eosinophilic esophagitis (EoE) activity in each participant. The VAS was a 100-mm horizontal line on which the right extreme (100) was labeled "worst possible disease activity" and the left (0) was labeled "no disease activity." Investigators were instructed to consider the line for the VAS as a continuum with their own opinion of extremes on either end. Investigators drew a vertical line at a point that best approximated the participant's current level of EoE disease activity. The investigator was to take into consideration how esophageal disease was impacting the participant's daily activities. The following instruction was given to the investigators: "Using the visual analog scale below, please mark a vertical line on the scale to indicate your assessment of EoE activity in this participant at this time." A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, 12 weeks after the start of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 18 | 17 | 19 | 16
scores on a scale | -38.9 (28.02) | -30.2 (27.11) | -39.3 (22.89) | -35.7 (28.49)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.4197, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Medium Dose; Test type: Superiority or Other; p = 0.9787, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs High Dose; Test type: Superiority or Other; p = 0.8987, ANCOVA — [p-value comment as in outcome 5, analysis 1]

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Budesonide
Description: On the day that pharmacokinetic (PK) blood samples were obtained, each participant delayed the morning dose of study medication until instructed to dose in the clinic. The sampling timepoints included pre-dose (0), and 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose. The lower limit of quantitation (LLOQ) for the analytical method was approximately 20 pg/mL in plasma using 0.2 mL of the sample. Because the PK analyses for the medium and high dose oral budesonide suspension (OBS) groups were based on plasma samples collected following administration of identical single doses of OBS, the data for the medium-dose group (OBS once-daily) and high-dose group (OBS twice-daily) were summarized together.
Time Frame: Week 2, 4, or 8, or at the Final Treatment Evaluation
Population: The Pharmacokinetic (PK) Set, defined as all participants in the safety analysis set who received oral budesonide suspension (OBS) and had sufficient PK samples to calculate PK parameters.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- 0.35 mg Dose: Participants 2 to 9 years old received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc), with a total daily dose of 0.35 mg.
- 0.50 mg Dose: Participants 10 to 18 years old received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc), with a total daily dose of 0.50 mg.
- 1.4 mg Dose: Participants 2 to 9 years old received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and either placebo or OBS 0.2 mg/ml after breakfast (qAM, pc), with a total daily dose of 1.4 mg (medium dose group) or 2.8 mg (high dose group).
- 2.0 mg Dose: Participants 10 to 18 years old received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and either placebo or OBS 0.2 mg/ml after breakfast (qAM, pc), with a total daily dose of 2.0 mg (medium dose group) or 4.0 mg (high dose group).
Arm/Group | 0.35 mg Dose | 0.50 mg Dose | 1.4 mg Dose | 2.0 mg Dose
Number analyzed (Participants) | 4 | 5 | 15 | 13
pg/mL | 492.0 (417.81) | 195.0 (64.37) | 1019.5 (670.18) | 958.4 (527.64)

11. Secondary Outcome: Time to Maximum (Tmax) And Half Maximum (T1/2) Plasma Concentration of Budesonide
Description: On the day that pharmacokinetic (PK) blood samples were obtained, each participant delayed the morning dose of study medication until instructed to dose in the clinic. The sampling timepoints included pre-dose (0), and 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose. The lower limit of quantitation (LLOQ) for the analytical method was approximately 20 pg/mL in plasma using 0.2 mL of the sample. Because the PK analyses for the medium and high dose oral budesonide suspension (OBS) groups were based on plasma samples collected following administration of identical single doses of OBS, the data for the medium-dose group (OBS once-daily) and high-dose group (OBS twice-daily) were summarized together. T1/2 is the time to terminal elimination half-life.
Time Frame: Week 2, 4, or 8, or at the Final Treatment Evaluation
Population: The PK Set, defined as all participants in the safety analysis set who received oral budesonide suspension (OBS) and had sufficient PK samples to calculate PK parameters.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 0.35 mg Dose | 0.50 mg Dose | 1.4 mg Dose | 2.0 mg Dose
Number analyzed (Participants) | 4 | 5 | 15 | 13
hours
  T1/2 | 3.288 (0.8265) | 3.398 (0.7841) | 3.472 (2.6753) | 3.528 (1.0223)
  Tmax | 0.68 (0.360) | 1.20 (0.447) | 0.93 (0.372) | 1.12 (0.546)

12. Secondary Outcome: Area Under The Plasma Concentration-Time Curve (AUC) of Budesonide From Time Zero to Time of The Last Measurable Concentration (AUC0-last)
Description: as for outcome 10
Time Frame: Week 2, 4, or 8, or at the Final Treatment Evaluation
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Groups:
- 0.35 mg Dose: Participants 2 to 9 years received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc), with a total daily dose of 0.35 mg.
- 0.50 mg Dose: Participants 10 to 18 years received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc), with a total daily dose of 0.50 mg.
- 2.0 mg Dose: Participants 10 to 18 years received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and either placebo or OBS 0.2 mg/ml after breakfast (qAM, pc), with a total daily dose of 2.0 mg (medium dose group) or 4.0 mg (high dose group).
Arm/Group | 0.35 mg Dose | 0.50 mg Dose | 1.4 mg Dose | 2.0 mg Dose
Number analyzed (Participants) | 4 | 5 | 15 | 13
hr*pg/mL | 1139.5 (800.84) | 743.8 (425.26) | 3259.3 (2109.37) | 3636.9 (1769.88)

13. Secondary Outcome: Percent of Participants With Potential Corticosteroid-Related Treatment-Emergent Adverse Events (TEAEs)
Description: Corticosteroid-Related TEAEs included candidiasis, oesophageal candidiasis, crying, psychomotor hyperactivity, aggression, anger, anxiety, conduct disorder, emotional disorder, insomnia, or mood altered mood. Corticosteroid-Related TEAEs were assessed systematically during the treatment and taper periods.
Time Frame: 15 weeks after the start of treatment
Population: The Safety Analysis Set, defined as all randomized participants who received at least one dose of double-blind study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 21 | 21 | 19 | 20
percentage of participants | 9.5 | 9.5 | 21.0 | 15.0

14. Secondary Outcome: Mean Change in Blood Pressure (BP) at End of Treatment
Description: BP was assessed for each treatment group at baseline and at each post-baseline visit including the final treatment evaluation.
Time Frame: Baseline, 12 weeks after the start of treatment
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 21 | 21 | 19 | 20
mmHg
  Systolic BP | -1.5 (14.74) | 1.8 (11.13) | 3.5 (8.20) | 8.0 (13.58)
  Diastolic BP | -3.1 (10.31) | 0.5 (8.89) | 3.1 (9.18) | 5.1 (8.83)

ADVERSE EVENTS:
Description: Adverse events are presented for the Safety Analysis Set, defined as all randomized participants who received at least one dose of double-blind study drug. Treatment group assignment was the treatment actually received. One participant in the medium dose group was enrolled and randomized then withdrew consent and did not receive study drug.
Groups:
- Low Dose: Participants received oral budesonide suspension (OBS) 0.05 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc) for 12 weeks with a 3 week taper period.
- Medium Dose: Participants received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and placebo after breakfast (qAM, pc) for 12 weeks with a 3 week taper period.
- High Dose: Participants received oral budesonide suspension (OBS) 0.2 mg/mL at bedtime (hs) and after breakfast (qAM, pc) for 12 weeks with a 3 week taper period.
Arm/Group | Placebo | Low Dose | Medium Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/19 | 1/20
Other Adverse Events (participants affected / at risk) | 10/21 | 13/21 | 16/19 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Low Dose (N=21) | Medium Dose (N=19) | High Dose (N=20)
Diet refusal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Low Dose (N=21) | Medium Dose (N=19) | High Dose (N=20)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 2 (2) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1) | 2 (3) | 2 (2) | 3 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (5) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 3 (4) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Crying (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Emotional Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early Satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.